CLINICAL TRIAL: NCT03446430
Title: Validation of Laser Doppler Vibrometer (LDV) for Measurement of Arterial Stiffness in Hypertensive Patients
Acronym: CARDIS-PWV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C17-43
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
Keywords: arterial stiffness; pulse wave velocity; laser Doppler vibrometry
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertensives (Experimental): PWV measurement by LDV
  Interventions: Device: PWV measurement by LDV

INTERVENTIONS:
Device: PWV measurement by LDV — PWV measurement by LDV : carotid-femoral, carotid and chest-carotid

SUMMARY:
The aim is to compare a new technique for assessing local and regional arterial stiffness: the Laser Doppler Vibrometry with the reference techniques, the applanation tonometry and echotracking.

DETAILED DESCRIPTION:
Cardiovascular (CV) diseases and their risk factors are the major contributors to global morbidity and mortality. CV diseases are responsible for over 17.3 million deaths per year worldwide, representing 30% of all global deaths. The measurement of arterial stiffness during the medical investigation of a hypertensive subject is essential to estimate the overall CV risk. The European Society of Hypertension (ESH) and the European Society of Cardiology (ESC) working group recommend its use for CV risk assessment. Indeed, arterial stiffness is currently the subject of a scientific consensus due to the large number of pathophysiological, epidemiological and pharmacological studies demonstrating that it integrates the duration and the level of exposure of the patient to known and identified CV risk factors (hypertension, tobacco, diabetes...) as well as those still discussed or more difficult to quantify (low birth weight, inflammation, infection, genetics...).

Arterial stiffness can be assessed in a number of ways, but the non-invasive measurement of the carotid-femoral pulse wave velocity (cfPWV) by applanation tonometry is regarded as the current gold standard because it corresponds to the aortic stiffness and it has been widely validated in epidemiological studies. However, the routine measurement of PWV by applanation tonometry is technically demanding and uncomfortable for the patient because the sensors can be attached around the neck or involve a palpation of the groin. The more advanced devices for PWV assessment are bulky, require trained operators due to the complexity of the procedure, and are relatively expensive. Therefore, none of the devices available for measurement of PWV are suitable for use in primary care. Measurement of arterial stiffness at primary care would allow large population screening for CV risks and thus enable more accurate CV risk prediction to better target preventive therapy among those individuals considered to be at low or moderate risk according to current guidelines. However, the tools and devices available today do not allow for mobile, low-cost, reliable, fast and non- or minimally-invasive point-of-care screening for measurement of arterial stiffness.

PWV measurement by laser Doppler vibrometry, contactless, is more comfortable, acceptable and could thus be a substitute for applanation tonometry.

A laser Doppler vibrometer (LDV) is an instrument that is used to make non-contact vibration measurements of a surface. The laser beam from the LDV is directed at the surface of interest (in our case the skin covering the artery or the heart), and the vibration amplitude and frequency are extracted from the Doppler shift of the reflected laser beam frequency due to the motion of the surface. Preliminary data suggest that LDV can lead to an improved screening and assessment of CV risk as a technique that makes it possible to measure aortic and local PWV. Indeed, Ghent University has successfully demonstrated that aortic PWV can be correctly measured with LDV. This method will greatly simplify procedures for measuring aortic stiffness if it is available in a compact form and adapted to clinical practice. This is the purpose of the CARDIS project, H2020 (http://www.cardis-h2020.eu/), which aims to develop a compact device for measuring local and segmental arterial stiffness without contact to the skin thanks to the LDV technique. The objective of this study is to compare the CARDIS LDV prototype with the reference techniques, carotid-femoral and local carotid PWV.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade I-III essential arterial hypertension, recently diagnosed, well controlled or insufficiently equilibrated under stable antihypertensive treatment for their HTA

Exclusion Criteria:

* Severe pathologies interfering with HTA or not allowing measurement by the techniques of interest, including skin diseases impeding the applanation tonometry
* Allergies to ultrasound gel or to adhesive film

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
carotid-femoral PWV measured by LDV | day 1

SECONDARY OUTCOMES:
carotid PWV measured by LDV | day 1
chest-carotid PWV measured by LDV | day 1
carotid-femoral PWV measured by applanation tonometry | day 1
carotid PWV measured by Echotracking | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Boutouyrie, MD, PhD, Principal Investigator — Pharmacology Department - Hopital Européen Georges Pompidou - Paris
Locations (1):
- Hopital Européen Georges Pompidou / Service de Pharmacologie, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker MA. Case of localized recombination in 23S rRNA genes from divergent bradyrhizobium lineages associated with neotropical legumes. Appl Environ Microbiol. 2001 May;67(5):2076-82. doi: 10.1128/AEM.67.5.2076-2082.2001. PMID 11319084
- [Derived] Badhwar S, Marais L, Khettab H, Poli F, Li Y, Segers P, Aasmul S, de Melis M, Baets R, Greenwald S, Bruno RM, Boutouyrie P. Clinical Validation of Carotid-Femoral Pulse Wave Velocity Measurement Using a Multi-Beam Laser Vibrometer: The CARDIS Study. Hypertension. 2024 Sep;81(9):1986-1995. doi: 10.1161/HYPERTENSIONAHA.124.22729. Epub 2024 Jun 27. PMID 38934112